CLINICAL TRIAL: NCT01772810
Title: A Phase 1, Open-label, Single-site, Safety Study of Human Spinal Cord-derived Neural Stem Cell Transplantation for the Treatment of Chronic SCI
Brief Title: Safety Study of Human Spinal Cord-derived Neural Stem Cell Transplantation for the Treatment of Chronic SCI
Acronym: SCI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neuralstem Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS2010-1
Record Dates: First submitted 2013-01-14; First posted 2013-01-21 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: Paralysis, spinal cord injury, chronic spinal cord injury, cspine injury, neck injury
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis; Neck Injuries | interventions — Creb3l2 protein, rat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgical implantation of human spinal cord stem cells (Experimental): Surgical implantation of human spinal cord derived neural stem cells.
  Interventions: Drug: Human spinal cord stem cells.

INTERVENTIONS:
Drug: Human spinal cord stem cells. — Human spinal cord stem cell implantation in paralysis patients due to a spinal cord injury.
  Other Names: spinal cord injury (SCI)

SUMMARY:
This is a safety study of human spinal cord-derived neural stem cell (HSSC) transplantation for the treatment of chronic spinal cord injury.

DETAILED DESCRIPTION:
Phase I, open-label, single-site, safety study of HSSC transplantation for the treatment of chronic spinal cord injury (SCI). Group A enrolled 4 subjects with a cord injury at T2-T12; Group B will enroll 4 subjects with a C5-C7 cord injury. Study period will be 6 months post-operative. Post-study, subjects will be followed for an additional 54 months.

ELIGIBILITY:
Inclusion Criteria:

* Lives within 500 miles of study center (For Group B)

  1. Have the ability to understand the requirements of the study, provide written informed consent, understand and provide written authorization for the use and disclosure of Protected Health Information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) Privacy Ruling] and comply with the study procedures
  2. Men and women 18-65 years old
  3. Women must have a negative serum pregnancy test and practice an acceptable method of contraception or be of non-childbearing potential (post-menopausal for at least 2 years or who have undergone hysterectomy or oophorectomy or surgical sterilization)
  4. At least 1 year but no more than 2 years from time of injury at the time of surgery
  5. SCI injury classified as AIS-A complete as confirmed by the PI and a Physical Medicine and Rehabilitation doctor or other SCI Medicine board certified physician based on a complete ISNC SCI examination
  6. Neurologic level of injury:

     1. Group A: injury within cord segments T2-T12;
     2. Group B: injury within cord segments C5-C7
  7. Confirmation of bone fusion by CT scan
  8. Agrees to the visit schedule as outlined in the informed consent
  9. All required vaccinations current at the time of enrollment: tetanus/diptheria (TDAP), herpes zoster/shingles (Zostavax®: within last 10 years and must be prior to surgery), pneumonia (Pneumovax®), seasonal/H1N1 flu vaccines (as appropriate for season). Any missing vaccination will be provided at the screening if consented by the otherwise eligible patient who will then be scheduled for surgery no less than 30 days post vaccination.

Exclusion Criteria:

1. SCI due to penetrating trauma such as gun shot or stabbing wound
2. SCI injuries involving complete spinal cord transection
3. Etiology of paraplegia or weakness related to other or additional neurologic process
4. MRI evidence of syrinx, multiple cysts, or a cyst with greater than 2cm in length or injury site involving greater than 2cm of the cord
5. Current or peak Panel Reactive Antibody (PRA) due to alloantibodies > 20% receiving their first allograft or presence of antibodies against HLA of the donor cells
6. Receipt of any investigational drug or device within 30 days prior to surgery
7. Receipt of any cell infusion other than blood transfusion
8. Any concomitant medical disease or condition noted below:

   1. Coagulopathy with INR > 1.4 at the time of screening
   2. Active infection
   3. Active hypotension requiring vasopressor therapy
   4. Skin breakdown over the site of surgery
   5. History of Malignancy (except for non-melanoma skin cancer)
   6. Primary or secondary immune deficiency
   7. Persistent MRI artifact that would prevent imaging post-op h. Creatinine >1.5, liver function tests (SGOT/SGPT, Bilirubin, Alk Phos) > 2x upper limit of normal, hematocrit/hemoglobin < 30/10, total WBC < 3000, uncontrolled hypertension (systolic > 180 or diastolic > 100) or uncontrolled diabetes (defined as hemoglobin A1C >8), evidence of GI bleeding by hemoccult test, positive tuberculosis, hepatitis B or C, or human immunodeficiency virus (HIV)
9. Presence of any of the following conditions:

   1. Current drug abuse or alcoholism
   2. Unstable medical conditions
   3. Unstable psychiatric illness including psychosis and untreated major depression
10. Any condition that the Investigator or primary physician feels may interfere with participation in the study
11. Any condition that the surgeon feels may pose complications for the surgery
12. Known hypersensitivity to basiliximab, tacrolimus or mycophenolate mofetil
13. Inability to provide informed consent as determined by screening protocol.
14. Stage III or above decubitus wound, other open wound, or active colostomy;
15. Autoimmune diseases, for which chronic corticosteroids or immunosuppression therapy may be needed;
16. Implanted spine stimulator;
17. Uncontrolled spasticity;
18. Uncontrolled neuropathic pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events and clinically significant laboratory abnormalities | 6 months

SECONDARY OUTCOMES:
Graft survival in the transplant site as determined by MRI (for Group A) and via autopsy, if one is completed. | Month 60
  Effectiveness of immunosuppression as determined by absence of donor-specific HLA antibodies.

OTHER OUTCOMES:
EMG, SCIM, ISNC SCI, and Bowel and bladder follow-up | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ciacci, MD, Principal Investigator — UCSD Medical Center, Division of Neurosurgery
Locations (1):
- UCSD Medical Center, Division of Neurosurgery, San Diego, California, United States

REFERENCES:
- [Derived] Martin JR, Cleary D, Abraham ME, Mendoza M, Cabrera B, Jamieson C, Marsala M, Ciacci JD. Long-term clinical and safety outcomes from a single-site phase 1 study of neural stem cell transplantation for chronic thoracic spinal cord injury. Cell Rep Med. 2024 Dec 17;5(12):101841. doi: 10.1016/j.xcrm.2024.101841. Epub 2024 Dec 2. PMID 39626671
- See also: Related Information — http://neuralstem.com